CLINICAL TRIAL: NCT05046925
Title: PACU or ICU for Postoperative Care After Major Thoracic and Abdominal Surgery：a Prospective Randomized Clinical Trial
Brief Title: PACU for Postoperative Care After Major Thoracic and Abdominal Surgery
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Responsible Party: Principal Investigator, xiangming fang, Director, Head of Anesthesiology and Critical Care, Principal Investigator, Professor, First Affiliated Hospital of Zhejiang University
Other Study IDs: PACU
Record Dates: First submitted 2021-09-04; First posted 2021-09-16 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-09

CONDITIONS: Anesthesia; Surgery--Complications
Keywords: Post-anesthetic care unit; Intensive care unit; Major surgery; postoperative complications; mortality; safety; efficacy; Postoperative care
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 24-hour PACU group: closely monitor in post-anesthetic unit (PACU) and the stay time is less than 24 hours, then patients can be discharged to floor
  Interventions: Procedure: postoperatively transferral to PACU
- 24-hour ICU group: closely monitor in intensive care unit (ICU) and the stay time is less than 24 hours, even patients die within 24 hours in ICU
  Interventions: Procedure: postoperatively transferral to ICU

INTERVENTIONS:
Procedure: postoperatively transferral to PACU — patients undergoing major thoracic and abdominal surgery will be transferred to PACU for postoperative care.
  Other Names: 24-hour PACU group
  Groups: 24-hour PACU group
Procedure: postoperatively transferral to ICU — patients undergoing major thoracic and abdominal surgery will be transferred to ICU for postoperative care.
  Other Names: 24-hour ICU group
  Groups: 24-hour ICU group

SUMMARY:
The aim of this study is to demonstrate the efficacy and safety of a specialised post-anaesthetic care unit (PACU) to a conventional intensive care unit (ICU) in adult patients after major thoracic and abdominal surgery. A better understanding of PACU for postoperative care is likely to reduce mortality and postoperative complications.

DETAILED DESCRIPTION:
With the continuous progress of surgical techniques, the number of major thoracic and abdominal surgeries is also increasing. Although intensive monitoring and initiative treatment benefit patients undergoing major surgery, there is also an increasing demand for intensive care in hospitals, which can lead to capacity limitations in the intensive care unit (ICU). In addition, there is emerging opinion that many patients after major thoracic and abdominal surgery do not require ICU care postoperatively to be provided safe and appropriate care. For hospitals and their staff the challenge is to optimize clinical processes and to optimize the effectiveness of treatment in regard to patient's outcome. Studying patient postoperative care following major thoracic and abdominal surgery exposes many opportunities to the improvement of patient safety, tailor the intensive care resource allocation and consider the costs and benefits of the options.

Postoperative mortality and morbidity remain major challenges, and most of these complications develop during the early postoperative period when patients have left the recovery room. Thus improving the care that patients receive once complications have occurred is crucial for reducing mortality. The post-anesthetic care unit (PACU) provides general to intensive care to immediate postsurgical patients. Patients with major thoracic and abdominal surgery surgeries are often kept in PACU until their condition is stabilized before shifting them to their designated wards or ICU[9]. Ender et al. and Probs et al. showed that treatment in a specialized PACU rather than an ICU, after cardiac surgery leads to earlier extubation, decreased ICU length of stay (LOS) and quicker discharge of hospital without compromising patient safety. Kastrup et al. described, introduction of a PACU staffed with intensivist coverage around the clock might shorten the hospital LOS and more patients can be treated in the same time, due to a better use of resources. Some other study described the transferral to a PACU as an unfavourable option, since equipment, expertise and staffing levels in the PACU are different from the ICU.

The possible solution to this problem might be the inclusion of the PACU in the process of distribution of patients to the different levels of intensive care for ensuring the timely recognition and effective management of postoperative complications in patients after major thoracic and abdominal surgery. The most challenges are to identify those candidates who can be monitored PACU within 24 hours postoperatively, rather than in ICU, and implement change in care paradigms safely.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years and older
* Undergoing major thoracic and abdominal surgery
* Postoperative hospital stay expected to be at least one night
* Patients requiring less than 24 hour stay in PACU or ICU

Exclusion Criteria:

* Patients aged less than 18 years
* Not receive major thoracic and abdominal surgery
* Stay in ICU is over 24 hours
* Hospital stay is less than 24 hours
* Patient not signing the informed consensus

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients undergoing major thoracic and abdominal surgery between September, 2021 and September, 2023 will be included in this study
Sampling Method: Probability Sample
Enrollment: 18000 (Estimated)
Dates: Start 2021-10-01 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
mortality | up to 90 days
  in-hospital mortality, 30-day and 90-day mortality

SECONDARY OUTCOMES:
Incidence of a composite of all-cause death, re-operation and major postoperative complications within 24 hours post surgery | within 24 hours postoperatively
  The primary outcome that will be measured is a composite of all-cause death, re-operation and major postoperative complications within 24 hours post surgery
The time of length of stay (LOS) | within 24 hours postoperatively
  LOS in PACU or ICU
incidence of care escalation | within 24 hours postoperatively
  patients in PACU is transferred to ICU within 24 hours rather than to floor
Incidence of major complications | 30 days postoperatively
  Postoperative major complications, defined by International Classification of Diseases, Tenth Revision (ICD-10) diagnostic codes
The time of hospital length of stay (LOS) | up to 30 days
  hospital length of stay (LOS)
medical cost | up to 90 days]
  Any medical cost during hospital stay
Incidence of emergency department (ED) visits | 90 days
  Emergency department (ED) visits within 90 days of the index surgery
Ventilation time | up 30 days
  Ventilation time postoperatively
Anaesthetic resuscitation time | Up to 24 hours
  Anaesthetic resuscitation time postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Xiangming Fang, Professor, Principal Investigator — First Affilated Hospital of Zhejiang University
Locations (1):
- First affilated hospital of zhejiang university, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided
Share all the data after the first article was published on issue

REFERENCES:
- [Result] International Surgical Outcomes Study group. Global patient outcomes after elective surgery: prospective cohort study in 27 low-, middle- and high-income countries. Br J Anaesth. 2016 Oct 31;117(5):601-609. doi: 10.1093/bja/aew316. PMID 27799174
- [Result] Weiser TG, Regenbogen SE, Thompson KD, Haynes AB, Lipsitz SR, Berry WR, Gawande AA. An estimation of the global volume of surgery: a modelling strategy based on available data. Lancet. 2008 Jul 12;372(9633):139-144. doi: 10.1016/S0140-6736(08)60878-8. Epub 2008 Jun 24. PMID 18582931
- [Result] Pastores SM, Kvetan V, Coopersmith CM, Farmer JC, Sessler C, Christman JW, D'Agostino R, Diaz-Gomez J, Gregg SR, Khan RA, Kapu AN, Masur H, Mehta G, Moore J, Oropello JM, Price K; Academic Leaders in Critical Care Medicine (ALCCM) Task Force of the Society of the Critical Care Medicine. Workforce, Workload, and Burnout Among Intensivists and Advanced Practice Providers: A Narrative Review. Crit Care Med. 2019 Apr;47(4):550-557. doi: 10.1097/CCM.0000000000003637. PMID 30688716
- [Result] Nates JL, Nunnally M, Kleinpell R, Blosser S, Goldner J, Birriel B, Fowler CS, Byrum D, Miles WS, Bailey H, Sprung CL. ICU Admission, Discharge, and Triage Guidelines: A Framework to Enhance Clinical Operations, Development of Institutional Policies, and Further Research. Crit Care Med. 2016 Aug;44(8):1553-602. doi: 10.1097/CCM.0000000000001856. PMID 27428118
- [Result] Loer SA. Anesthesiologists should bring in their expertise during the early postoperative period to improve surgical outcome. Curr Opin Anaesthesiol. 2018 Dec;31(6):713-715. doi: 10.1097/ACO.0000000000000663. No abstract available. PMID 30247164
- [Result] Lalani SB, Ali F, Kanji Z. Prolonged-stay patients in the PACU: a review of the literature. J Perianesth Nurs. 2013 Jun;28(3):151-5. doi: 10.1016/j.jopan.2012.06.009. PMID 23711311
- [Result] Kellner DB, Urman RD, Greenberg P, Brovman EY. Analysis of adverse outcomes in the post-anesthesia care unit based on anesthesia liability data. J Clin Anesth. 2018 Nov;50:48-56. doi: 10.1016/j.jclinane.2018.06.038. Epub 2018 Jun 29. PMID 29979999
- [Result] Belcher AW, Leung S, Cohen B, Yang D, Mascha EJ, Turan A, Saager L, Ruetzler K. Incidence of complications in the post-anesthesia care unit and associated healthcare utilization in patients undergoing non-cardiac surgery requiring neuromuscular blockade 2005-2013: A single center study. J Clin Anesth. 2017 Dec;43:33-38. doi: 10.1016/j.jclinane.2017.09.005. Epub 2017 Sep 30. PMID 28972924
- [Result] Probst S, Cech C, Haentschel D, Scholz M, Ender J. A specialized post anaesthetic care unit improves fast-track management in cardiac surgery: a prospective randomized trial. Crit Care. 2014 Aug 15;18(4):468. doi: 10.1186/s13054-014-0468-2. PMID 25123092
- [Result] Ender J, Borger MA, Scholz M, Funkat AK, Anwar N, Sommer M, Mohr FW, Fassl J. Cardiac surgery fast-track treatment in a postanesthetic care unit: six-month results of the Leipzig fast-track concept. Anesthesiology. 2008 Jul;109(1):61-6. doi: 10.1097/ALN.0b013e31817881b3. PMID 18580173
- [Result] Kastrup M, Seeling M, Barthel S, Bloch A, le Claire M, Spies C, Scheller M, Braun J. Effects of intensivist coverage in a post-anaesthesia care unit on surgical patients' case mix and characteristics of the intensive care unit. Crit Care. 2012 Jul 18;16(4):R126. doi: 10.1186/cc11428. PMID 22809294
- [Result] Duke GJ. Metropolitan audit of appropriate referrals refused admission to intensive care. Anaesth Intensive Care. 2004 Oct;32(5):702-6. doi: 10.1177/0310057X0403200518. PMID 15535499